CLINICAL TRIAL: NCT06832462
Title: The Efficacy of a One-Day Acceptance and Commitment Therapy in Enhancing Mental Health and Psychological Capital Among University Students.
Brief Title: A Prospective and Experimental Study on Efficacy of One-Day of Acceptance and Commitment Therapy on Mental Health Among University Students. a Psychological Capital Examine As Mediator to the Efficacy of ACT on Mental Health.
Acronym: ACT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Teknologi Malaysia (Other)
Responsible Party: Principal Investigator, Akmar Nabila Binti A Bakar, Postgraduate Student, Universiti Teknologi Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UTMREC-2024-83; Q.J130000.3853.31J93 (Other Grant/Funding Number: UTMER)
Record Dates: First submitted 2025-02-13; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Mental Health (Depression); Mental Health Issues; Anxiety
Keywords: Acceptance and Commitment Therapy (ACT); University student; Animation video efficacy
MeSH Terms: conditions — Psychological Well-Being; Depression; Anxiety Disorders | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: There are two group: intervention and waitlist (control)
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): This group will receive one-day Acceptance and Commitment Therapy (ACT). The therapy include 4 sessions that explain and guide participants to understand the concept of ACT and apply in their daily life for the purpose of enhancing good mental health.
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Waitlist Group (Other): After one month, the waitlist group will receive the same intervention to ensure the result of efficacy of one-day acceptance and commitment therapy (ACT) in the intervention group can be compared with the waitlist group.
  Interventions: Behavioral: Acceptance and Commitment Therapy

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — A one-day Acceptance and Commitment Therapy (ACT) will be held with three (3) sessions. The sessions start with ice breaking, and follow by,
  The first session will build a therapeutic relationship and icebreaking, using animated video (unwanted guest) presentations to explain how ACT can help manage issues.
  The second session will focus on acceptance and defusion concepts, emphasizing the importance of letting go of unproductive emotion-control techniques by using animated video (response ability)
  The third session, 'Show Up', will increase awareness of undesirable thoughts and feelings through structured mindfulness exercises and observing surroundings. The therapist will explain the metaphor of dropping the anchor and emphasize the

SUMMARY:
This prospective and experimental study examines the efficacy and feasibility of a one-day ACT intervention on mental health, psychological flexibility, and psychological capital among university students. Other than that, this study examines the mediator role of psychological capital in the mechanism through which Acceptance and Commitment Therapy (ACT) improves mental health issues among university students. Animation video efficacy will be examined to determine whether it helps in enhancing students' understanding of Acceptance and Commitment Therapy (ACT).

The main questions it aims to answer are:-

1. What are the correlation between psychological capital, psychological flexibility, depression and anxiety?
2. How does one-day ACT intervention affect mental health (depression and anxiety) and psychological capital among university students?
3. Does psychological capital mediate the effect of psychological flexibility on mental health issues among university students
4. Do video presentations improve the understanding of ACT concepts?
5. Is one-day ACT intervention feasible to be implemented among university students?

Researchers will compare to see if there are any differences between the intervention group and waitlist groups of university students' levels of depression, anxiety, psychological flexibility and psychological capital.

Participants will:

* Participate in a one-day Acceptance and Commitment Therapy (ACT) intervention.
* Answer questionnaires at four (4) different phases.
* Follow up after one month and answer survey questions about the effect of ACT on their mental health level.

DETAILED DESCRIPTION:
This is a prospective and experimental study. A prospective study approach is used to examine the changes in outcome measures along with the data collection timeline. Data will be collected at four different points: screening (T1), pre-intervention (T2), post-intervention (T3), and one month after intervention (T4). This is an experimental study, a randomized control trials study, and consists of two arms: a one-day ACT intervention and waitlist groups. The efficacy of a one-day ACT intervention will be evaluated using a randomized controlled trial approach by comparing the differences between intervention and waiting groups.

This is a prospective and experimental study. A prospective study approach is used to examine the changes in outcome measures along with the data collection timeline.

Data will be collected at four different points: screening (T1), pre-intervention (T2), post-intervention (T3), and one month after intervention (T4).

This is an experimental study, a randomized control trials study, and consists of two arms: a one-day ACT intervention and waitlist groups. The efficacy of a one-day ACT intervention will be evaluated using a randomized controlled trial approach by comparing the differences between intervention and waiting groups.

(T1) - Preliminary phase - A set of questionnaires of the Beck Anxiety Inventory (BAI) and Beck Depression Inventory (BDI) will be distributed through the student portal for screening. Potential participants who score moderate and above will be invited to the One-Day ACT intervention. The details of potential participants will be recorded.

(T2) - During pre-intervention, participants will be divided into two groups: a waitlist and a group that will receive batteries of questionnaires. The questionnaires included the demographic survey, BAI, BDI, Acceptance and Action Questionnaire II (AAQ-II) and Psychological Capital Questionnaires (PCQ) to participants before receiving ACT intervention. Those who answer the questionnaires will receive a One-Day ACT intervention. In addition, respondents will be fully informed regarding the objectives and procedure of this research, and consent information will be gathered.

One-Day Intervention: -

A one-day ACT intervention will be conducted in three sessions, each lasting 40 minutes. The intervention is based on a module developed by Shari et al. (2020) and aims to help respondents manage their issues, such as unpleasant thoughts and feelings.

The first session will build a therapeutic relationship and icebreaking, using animated video (unwanted guest) presentations to explain how ACT can help manage issues.

The second session will focus on acceptance and defusion concepts, emphasizing the importance of letting go of unproductive emotion-control techniques by using animated video (response ability)

The third session, 'Show Up', will increase awareness of undesirable thoughts and feelings through structured mindfulness exercises and observing surroundings. The therapist will explain the metaphor of dropping the anchor and emphasize the importance of being present and aware of oneself.

The final session, 'Get Moving', will connect values to practical action plans, using animated video (Values VS Goals) presentations to help respondents define their values and identify significant life steps.

(T3) - post-intervention, where a one-day ACT intervention has been done and a set of questionnaires distributed to participants. The questionnaires include BAI, BDI, AAQ-II, PCQ, and Treatment satisfaction questionnaire and Learner Acceptance scale will be used to measure the effectiveness of video presentation used during intervention.

(T4) - After one month of intervention, this phase will follow up with the participants who undergo One-Day ACT intervention by answering BAI, BDI, AAQ-II and PCQ questionnaires.

All data collected will be analysed using SPSS 26 to examine the research objective and hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Local Malaysian Students
* 18 years old and above
* Students who score moderate and above for Beck Depression Inventory (BDI) and Beck Anxiety Inventory (BAI) during screening phase.

Exclusion Criteria:

* International students
* Those who received or are undergoing Acceptance and Commitment Therapy (ACT)
* Those who have psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
A one-day ACT intervention is effective in enhancing mental health | Before and after participate the one-day acceptance and commitment therapy.
  The efficacy of ACT on mental health among university student will be measure by using Beck anxiety and Beck Depression Inventory pre and post of the intervention between intervention and waitlist group. We will compare the result (changes) between pre-intervention and post-intervention between waitlist and intervention. Effect size also will be calculated.

SECONDARY OUTCOMES:
Psychological capital and psychological flexibility. | Before and after participate the one-day acceptance and commitment therapy.
  Psychological capital will be measured using the Psychological Capital Questionnaire (PCQ). Meanwhile Psychological flexibility is measured by using the Acceptance and action questionnaire (AAQ II)
Psychological flexibility mediates the mechanism through which ACT improves mental health issues among university students. | Before and after participate the one-day acceptance and commitment therapy.
  Mediation analysis is calculated by using PROCESS macro Version 3.5 developed by Andrew F. Hayes. Single mediator model will be used to analyse total, direct, and indirect effect of the mediator variables

OTHER OUTCOMES:
Video presentations are effective in improving understanding of the ACT concepts. | Before and after participate the one-day acceptance and commitment therapy.
  The score from the survey of The Learning Acceptance Scale will be calculated to determine the efficacy of video presentations in enhancing the understanding of ACT concepts. The score is...
A one-day ACT intervention is feasible to be implemented in enhancing mental health and psychological capital among university students | After participate a one-day acceptance and commitment therapy
  The score for The Treatment Satisfaction Questionnaire and at T3 will be computed into the total score to determine the level of satisfaction toward the therapy and the therapist.

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Teknologi Malaysia, Johor Bahru, Johor, Malaysia

IPD SHARING:
Plan to Share IPD: No
In the inform consent, we agreed to keep the information private and confidential.